CLINICAL TRIAL: NCT05468944
Title: Robotic Transanal Specimen Extraction Surgery Versus Robotic Transabdominal Incision Specimen Extraction Surgery for Patients With Rectal Cancer: A Multicenter Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taiyuan Li (Other)
Responsible Party: Sponsor-Investigator, Taiyuan Li, Professor, The First Affiliated Hospital of Nanchang University
Organization: The First Affiliated Hospital of Nanchang University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RO220624
Record Dates: First submitted 2022-07-13; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Rectal Neoplasms; Robotic Surgery; Natural Orifice Specimen Extraction Surgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transanal group (Experimental): Participants in this group underwent robotic surgery with transanal specimen extraction
  Interventions: Procedure: Transanal specimen extraction robotic surgery
- Transabdominal group (Active Comparator): Participants in this group underwent robotic surgery with transabdominal specimen extraction
  Interventions: Procedure: Transabdominal specimen extraction robotic surgery

INTERVENTIONS:
Procedure: Transanal specimen extraction robotic surgery — Participants in this group underwent robotic rectal cancer resection ,the specimens were extracted through anus.
  Arms: Transanal group
Procedure: Transabdominal specimen extraction robotic surgery — Participants in this group underwent robotic assisted rectal cancer resection ,the specimens were extracted through the incision on the abdominal wall.
  Arms: Transabdominal group

SUMMARY:
This prospective, multicenter, randomized, open-label study aims to evaluate the perioperative safety and feasibility of specimen extraction through anus regarding robotic radical excision of rectal cancer.

DETAILED DESCRIPTION:
In this study, investigators will evaluate the perioperative safety and feasibility of robotic transanal specimen extraction surgery with robotic transabdominal incision specimen extraction surgery as a control.The study is prospective, randomized, open-label, and multicenter conducted at 12 centers. Considering the significance level and abscission rate, it is expected that a total of 556 subjects will be included in the two groups from January 2023 to June 2024, with the incidence of postoperative complications as the main study endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 75 years;
2. Historically confirmed rectal adenocarcinoma;
3. Diagnosed with rectal cancer by pelvic/rectal magnetic resonance imaging;
4. cT1-4aNxM0 high rectal adenocarcinoma; cT1-3NxM0 mid/low rectal adenocarcinoma;
5. No evidence of distant metastases;
6. A maximum of 5cm in diameter;
7. Body mass index (BMI) ≤ 30 kg / m2;
8. No local complications (no obstruction, incomplete obstruction, no massive active bleeding, no perforation, preoperatively abscess formation, no local invasion);
9. Willing to undergo surgery;
10. Sign the informed consent;

Exclusion Criteria:

1. Presence of lateral/inguinal lymph node metastases;
2. Previous history of malignant colorectal tumor;
3. Multiple primary colorectal tumors;
4. Neoadjuvant therapy;
5. Salvage surgery for endoscopic surgery;
6. History of previous abdominopelvic surgeries or extensive intra-abdominal adhesion;
7. Familial adenomatous polyposis, Lynch syndrome, and inflammatory bowel disease;
8. Comorbid with other malignancies within 5 years;
9. ASA ≥ IV and/or ECOG performance status score ≥ 2;
10. Severe liver, kidney, cardiopulmonary insufficiency, coagulopathy or serious underlying diseases;
11. Serious mental illness;
12. Pregnant or lactating women;
13. Uncontrolled infection;
14. Abnormal anal function or anal stenosis;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Complication rate | Up to 30 days postoperatively.
  Complication rate within 1 month postoperatively.All complications of surgery will be documented and graded by the Clavien-Dindo classification system,generally including anastomotic leakage, abdominal infection, bleeding, incision infection, incision implantation, intestinal obstruction, and rectovaginal fistula.

SECONDARY OUTCOMES:
C-reactive protein (CRP) | 1 day before operation, 1, 3, 5 days postoperatively, and up to 2 weeks.
  Detection of serum CRP levels (mg/L) to evaluate surgical stress response and immune function.
Interleukin | 1 day before operation, 1, 3, 5 days postoperatively, and up to 2 weeks.
  Detection of serum levels of Interleukin-1 (IL-1), interleukin-6 (IL-6), interleukin-8 (IL-8), interleukin-10 (IL-10) (pg/L) to evaluate surgical stress response and immune function.
Cortisol | 1 day before operation, 1, 3, 5 days postoperatively, and up to 2 weeks.
  Detection of Serum Cortisol Level (nmol/L) to evaluate surgical stress response and immune function.
CD3, CD4, and CD8 lymphocyte subsets | 1 day before operation, 1, 3, 5 days postoperatively, and up to 2 weeks.
  Count CD3, CD4, and CD8 lymphocyte subsets (pieces/ul) to assess surgical stress response and immune function.
Positive rate of tumor cells | Intraoperative.
  Intraoperative peritoneal lavage fluid will be collected both for aerobic culture and centrifuged ,stained and viewed to find exfoliated cancer cells.The sample will be considered positive if at least one tumor cell was detected.
bacterial positive rate | Intraoperative.
  Intraoperative peritoneal lavage fluid will be collected both for aerobic culture and centrifuged ,stained and viewed to find exfoliated cancer cells.The sample will be considered positive if at least one tumor cell was detected.
Pain assessment | 1 day before operation, 1, 2, 3 days postoperatively, and up to 2 weeks.
  Visual analogue scale (VAS) will be used to evaluate the postoperative pain. If analgesics were needed, the type and dose of analgesics after operation should be recorded.
Wexner scale | 1 day before operation, and 1, 3, 6 months postoperatively.
  Wexner scale (0 are normal continence, 20 are maximum incontinence with maximum disturbance of lifestyle) will be used to evaluate the defecation function.
LARS scale | 1 day before operation, and 1, 3, 6 months postoperatively.
  LARS scale(0~20 points are defined as no LARS, Scores from 21 to 29 were defined as mild LARS, and from 30 to 42 as severe LARS. The higher the score, the worse the anal bowel function) will be used to evaluate the defecation function.
Postoperative recovery composite | Up to 2 weeks.
  Including the time to first flatus (record the patient's first self induced exhaust time after operation, accurate to hours, and perform auscultation of bowel sounds regularly every day after operation), the time to first ambulation (hours), the time to first eating (hours) and the time to first defecation (hours).
EORTC QLQ-C30 | 1 day before operation, 1, 3, 6 months postoperatively.
  To assess the quality of life of all cancer patients.
EORTC QLQ-C38 | 1 day before operation, 1, 3, 6 months postoperatively.
  To assess the quality of life in patients with rectal cancer.
Tumor size | Up to 30 days postoperatively.
  To assess the quality of surgical specimens.
Number of Histopathological type | Up to 30 days postoperatively.
  To assess the quality of surgical specimens and postoperative pathological evaluation.
Degree of differentiation | Up to 30 days postoperatively.
  To assess the quality of surgical specimens and postoperative pathological evaluation.
Distance , positive condition of pathological margin (proximal, distal, circumferential) | Up to 30 days postoperatively.
  To assess the quality of surgical specimens and postoperative pathological evaluation.
Number of lymph node dissection and metastasis | Up to 30 days postoperatively.
  To assess the quality of surgical specimens and postoperative pathological evaluation.
Nerve vessel involvement rate | Up to 30 days postoperatively.
  To assess the quality of surgical specimens and postoperative pathological evaluation.
Hospitalization costs | Up to 30 days.
  To assess the financial burden difference.
Local recurrence rate | 1, 3, 5 years postoperatively.
  To assess the long-term postoperative outcomes.
The incidence rate of distant metastasis | 1, 3, 5 years postoperatively.
  To assess the long-term postoperative outcomes.
Tumor-free survival rates | 1, 3, 5 years postoperatively.
  To assess the long-term postoperative outcomes.
Overall survival rate | 1, 3, 5 years postoperatively.
  To assess the long-term postoperative outcomes.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing
  - The Second Xiangya Hospital, Central South University, Changsha
  - Three Gorges Hospital Affiliated to Chongqing University, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - The First Affiliated Hospital of Gannan Medical University, Ganzhou
  - The Second Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - The Second Affiliated Hospital of Harbin Medical University, Harbin
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Zhongshan Hospital, Fudan University, Shanghai
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Zhongshan Hospital of Xiamen University, Xiamen
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou